CLINICAL TRIAL: NCT05582252
Title: The Comprehensive Investigation to Define a New Scoring System for ICD Implantation Based on Genotypic and Phenotypic Criteria; A Multidisciplinary and Multicentral Genome-Wide Association Study
Brief Title: Genome-Wide Association Study With the Aim of Implantable Cardioverter Defibrillator Implantation Genophenotypic Risk Stratification
Acronym: ICDGPSS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Selcuk University (Other)
Collaborators: Ankara University (Other); TC Erciyes University (Other); Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ebru Marzioglu Ozdemir, Assistant Professor. Dr., Selcuk University
Other Study IDs: KINASK-ICDGPSS-EICCG2210; DN2022/400-MN2022/17 (Other: REPUBLIC OF TURKEY DEANARY OF SELCUK UNIVERSITY FACULTY OF MEDICINE)
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: ICD; Arrythmia; Sudden Cardiac Death
Keywords: Implantable Cardioverter Defibrillators; Ventricular Arrhythmia; Sudden Cardiac Death; Cardiogenomics; Cardiogenetics; GWAS; Genetic Polymorphism
MeSH Terms: conditions — Arrhythmias, Cardiac; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA extraction will be done following non-invasive saliva sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Experimental group: Patients with ICD who received at least one electric shock in 6 months after ICD implantation
  Interventions: Other: Non-Invasive saliva sampling
- Control Group: Patients with ICD who didnot received any electric shock in 6 months after ICD implantation
  Interventions: Other: Non-Invasive saliva sampling
- Healthy Group: Healthy Volunteers This group will be used for related bioinformatic analysis (DATA analysis stage) but not in statistical analysis
  Interventions: Other: Non-Invasive saliva sampling

INTERVENTIONS:
Other: Non-Invasive saliva sampling — There are two types of intervention in this ambidirectional study.
  1. Non-Invasive Saliva Sampling will be done for DNA extraction for the purpose of genetic analysis. This would be the prospective sampling and it's not part of the related medical centre's clinical routine.
  2. ICD that is already implanted in the patients and had been indicated by related medical centre's clinical routine approach. This is not a prospective approach to this study since the study would be retrospectively gathered phenotypic parameters from the hospital data records.
  Other Names: ICD

SUMMARY:
This clinical study will be conducted with funding from European Innovation Council(EIC) after approval of the fund grant and is part of our organization's European Pathfinder Project(Ref: HORIZON-EIC-2022-PATHFINDERCHALLENGES-01). The clinical study step of this project will be started in a retrospective time prospective manner by gathering the phenotypic(clinical measuring factors) data from patients who underwent ICD implantation therapy. The study will be done as a case-control type in which patients who did not get any shocks in 6 months post-implantation will be allocated to the control group. A customized and highly specific cardiogenomics panel will be designed and ordered to be specially manufactured as a standard kit by Illumina® (San Diego, California, U.S.) following an exhaustive investigation for collecting genetic variants which correlated to cardiovascular development. Mentioned kit bears the standard and validated technology which is part of the genetic tests routine and is being produced by Illumina® incorporate. However, as an option manufacturer is designing custom kits for research purposes by getting the desired variant lists using the same technology. Accordingly, enrolled patients in the study will be prospectively sampled ( Non-Invasive saliva sampling) for getting genetically analysed by Illumina®'s Infinium Assay Microarray platform with fully customized 700,000 single nucleotide polymorphism kits. The result of this sampling will be data and statistically analysed in a genome-wide association study(GWAS) manner by considering the 5x10-8 p.value and will be associated with each phenotypic parameter. Accordingly, the study will assess the genetic risk stratification in ICD patients in a much more detailed fashion. Following this assessment genophenotypic statistical analysed will be done to combine both parameters and generate a formula for scoring the indicator factors based on each odds ratio. Correspondingly, this new scaling formula will be analysed, verified and validated further by a randomized sampling of the population in our study before being stated. Additionally, This study will not only help to improve current genetic polymorphism clinal significant status (pathogenicity and significance of variant) but also can associate new markers with high significance that can be directly used in clinical screening, diagnosis or clinical approaches.

ELIGIBILITY:
Inclusion Criteria:

* ICD-implanted patients (both for primary and secondary intervention)
* Being a volunteer for the study
* Adequacy in understanding the study risks and accepting the Informed Consent Form
* Official acceptance of the legal and official parents (both father and mother), If younger than 18 years old

Exclusion Criteria:

* The patient who does not volunteer to involve to the study.
* Diagnosis of underlying arrhythmogenic disease (Structural Heart disease, Brugada, Arrhythmogenic right ventricular dysplasia, etc.)
* Development of electric shock due to acute coronary syndrome
* Atrial Fibrillation (AFib) With Rapid Ventricular Response
* Electric shock in patients with electrolyte imbalance-induced VT/VF
* Electric Shock in a patient with acute myocarditis-induced ventricular arrhythmias
* Patients that had an electric shock because of pacing / ATP ramp-induced VT (RV/CRT Pacing)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population are the ICD-implanted patients according to exclusion and inclusion criteria. No randomization will be done for patient selection and group allocation (the validation stage will be done by randomization). An extra-healthy volunteer will be included for bioinformatic data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Revealing SNP variants related to phenotypic measurement factors | 2024MAY
  ICD Shock, Sudden Cardiac Death, Ventricular Arrythmia and ICD prognosis related genetic polymorphism variant
GENOPHENOTYPIC risk stratification | 2024DEC
  Results of genotype and phenotype statistical analysis
Comprehensive genophenotypic scoring system formula | 2025MARCH
  a formula that is based on genetic and phenotypic parameters that can be used as criteria for ICD implantation indication

SECONDARY OUTCOMES:
offering a comprehensive cardiogenetic kit | 2025MARCH
  a kit that is based on the Illumina bead chip Infinium Microarray technology and can be used for research, clinical screening and diagnosis

OTHER OUTCOMES:
comprehensive local demographic statistics | 2024DEC
  since a large-scale study is desired, valuable domestic demographic statistical data can be achieved

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Genetic Department Faculty of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No